CLINICAL TRIAL: NCT02781038
Title: Smoking Cessation and a Teachable Moment in Patients With Acute Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 819551
Record Dates: First submitted 2016-05-02; First posted 2016-05-24 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Tobacco Use Disorder; Bone Fractures
MeSH Terms: conditions — Tobacco Use Disorder; Fractures, Bone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventional (Experimental): All subjects will receive a baseline attitude survey. At some point in their hospitalization, preferably at least one day later and no greater than one week later, the patients will be given a teaching intervention and receive another attitude survey.
  Interventions: Behavioral: Teaching intervention
- Control (Other): All subjects will receive a baseline attitude survey. At some point in their hospitalization, preferably at least one day later and no greater than one week later, the patients will receive another attitude survey.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Teaching intervention — Subjects will receive a pamphlet which describes the relationship between smoking and negative outcomes in fracture healing.
  Other Names: Pamphlet
  Arms: Interventional
Behavioral: Control — Subjects in this group will not receive the pamphlet
  Arms: Control

SUMMARY:
Patients who smoke and suffer from fractures are worse off than those who do not smoke. Orthopaedic patients represent a group that can benefit from physician contributions to smoking cessation, and a special opportunity to cue this can begin with the orthopaedic surgeon in the acute setting. However, the best way to appropriately counsel these patients and assess the impact as a teachable moment remains undetermined.

DETAILED DESCRIPTION:
If the patient self-identifies as a smoker, the investigators will consent and randomize to receive the intervention or not. Either way, all will receive a baseline attitude survey. The patient will be given a series of questions that target the areas of interest noted in the model. At some point in their hospitalization, preferably at least one day later and no greater than one week later, the patients will be given the teaching intervention (or not), and receive another attitude survey. After discharge, the patients will be expected in orthopaedic follow up clinic. At that time they will receive another attitude survey. If unable to deliver at that time, they will be contacted by phone or sought at their second clinic follow up.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 or over, who are not under the jurisdiction of the department of corrections
* Individuals receiving care from University of Pennsylvania Health System clinicians for orthopaedic injuries
* Individuals who self-identify as smokers

Exclusion Criteria:

* Under age 18
* Under the jurisdiction of the department of corrections
* Nonsmokers
* People not currently receiving fracture care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Attitude adjustment | Change from baseline (inpatient) pre-intervention, to 24 hours post-intervention, to first clinical follow up visit (outpatient) 1-3 weeks post-intervention
  Study-specific 9 question Likert-scale survey

SECONDARY OUTCOMES:
Exploratory Impact Assessment | Change from baseline (inpatient) pre-intervention, to 24 hours post-intervention, to first clinical follow up visit (outpatient) 1-3 weeks post-intervention
  Single binary question

CONTACTS AND LOCATIONS:
Overall Officials: Jaimo Ahn, MD, PhD, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Hadithy N, Sewell MD, Bhavikatti M, Gikas PD. The effect of smoking on fracture healing and on various orthopaedic procedures. Acta Orthop Belg. 2012 Jun;78(3):285-90. PMID 22822565
- [Background] Patel RA, Wilson RF, Patel PA, Palmer RM. The effect of smoking on bone healing: A systematic review. Bone Joint Res. 2013 Jun 14;2(6):102-11. doi: 10.1302/2046-3758.26.2000142. Print 2013. PMID 23836474
- [Background] An LC, Foldes SS, Alesci NL, Bluhm JH, Bland PC, Davern ME, Schillo BA, Ahluwalia JS, Manley MW. The impact of smoking-cessation intervention by multiple health professionals. Am J Prev Med. 2008 Jan;34(1):54-60. doi: 10.1016/j.amepre.2007.09.019. PMID 18083451
- [Background] Prochaska JO, DiClemente CC, Norcross JC. In search of how people change. Applications to addictive behaviors. Am Psychol. 1992 Sep;47(9):1102-14. doi: 10.1037//0003-066x.47.9.1102. PMID 1329589
- [Background] Lawson PJ, Flocke SA. Teachable moments for health behavior change: a concept analysis. Patient Educ Couns. 2009 Jul;76(1):25-30. doi: 10.1016/j.pec.2008.11.002. Epub 2008 Dec 24. PMID 19110395
- [Background] Fonarow GC. In-hospital initiation of statins: taking advantage of the 'teachable moment'. Cleve Clin J Med. 2003 Jun;70(6):502, 504-6. doi: 10.3949/ccjm.70.6.502. No abstract available. PMID 12828221
- [Background] Glasgow RE, Stevens VJ, Vogt TM, Mullooly JP, Lichtenstein E. Changes in smoking associated with hospitalization: quit rates, predictive variables, and intervention implications. Am J Health Promot. 1991 Sep-Oct;6(1):24-9. doi: 10.4278/0890-1171-6.1.24. PMID 10148681
- [Background] McBride CM, Emmons KM, Lipkus IM. Understanding the potential of teachable moments: the case of smoking cessation. Health Educ Res. 2003 Apr;18(2):156-70. doi: 10.1093/her/18.2.156. PMID 12729175
- [Background] Dohnke B, Ziemann C, Will KE, Weiss-Gerlach E, Spies CD. Do hospital treatments represent a 'teachable moment' for quitting smoking? A study from a stage-theoretical perspective. Psychol Health. 2012;27(11):1291-307. doi: 10.1080/08870446.2012.672649. Epub 2012 Apr 4. PMID 22472171